CLINICAL TRIAL: NCT05635682
Title: Investigation of the Relationship Between Sensation, Balance, Gait, Posture and Reaction Time in Individuals in Opioid Maintenance Treatment Process
Brief Title: Investigation of the Relationship Between Different Assesments in Individuals in Opioid Maintenance Treatment Process
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ilke Keser, Prof. Dr., Gazi University
Other Study IDs: 66442466-604.01.02
Record Dates: First submitted 2022-10-27; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Opioid Use Disorder
Keywords: opioid use disorder; plantar sensation; reaction time; balance; gait
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Study Group: Individuals in the process of maintenance therapy with opioid use disorder
  Interventions: Other: Observational and anthropometric assesments
- Control Group: Healty people
  Interventions: Other: Observational and anthropometric assesments

INTERVENTIONS:
Other: Observational and anthropometric assesments — Plantar sensation, foot reaction time, head and trunk proprioceptions, posture, balance and gait assesments

SUMMARY:
Opioid use disorder is the chronic use of opioids that causes clinically significant distress or impairment. More than 16 million people world wide are opioid addicts. The diagnosis of opioid use disorder is based on the Diagnostic and Statistical Manual of Mental Disorders (DSM-5). Despite the social and personal consequences of opioid use disorder in individuals; It consists of an excessive desire to use opioids, increased opioid tolerance, and withdrawal syndrome when discontinued. Examples of opioids include heroin, morphine, codeine, synthetic opioids such as fentanyl and oxycodone.

In many countries, the main pharmacological approach in the treatment of opioid use disorder is maintenance therapy using opioid agonists. The combination of buprenorphine and naloxone is one of the most effective agents used in maintenance therapy. Due to the effects of both opioid use and maintenance therapy, these individuals have sensory problems, balance and gait disturbances, and a prolonged reaction time.

The aim of this study is to examine the relationship between sensation, balance, gait, posture and reaction time in individuals on opioid maintenance therapy and to compare them with healthy individuals.

DETAILED DESCRIPTION:
This study will be conducted with the participation of 80 people between the ages of 18 and 65, including 40 individuals who have voluntarily agreed to participate in the study, who have received opioid use disorder according to the DSM V diagnostic criteria and are in the process of maintenance treatment, and 40 healthy individuals. Dec.

Within the scope of the study, the cognitive levels of the participants will be evaluated by Montreal Cognitive Assessment (MoCA).

Sensory evaluations will be made in the form of proprioception sense, light touch sense, vibration sense and two-point discrimination assessment. Proprioception assessments will be performed using a digital inclinometer for the neck and torso separately (J-Tech Dualer IQ, J-Tech Medical Industries, Salt Lake City, USA).

The posture assessment will be performed by the New York Posture Analysis Method.

The Semmes Weinstein Monofilament Test (SWMT) will be used to assess the sense of touch and pressure on the sole of the foot.The test will be applied to the first metatarsal head, medial foot, lateral foot and heel. 3 Repetitions will be performed for each zone. At the end of the test, the values of the four regions will be added and divided into four and the average value will be calculated. The right and left extremities will be evaluated separately.

A 128 Hz diaposon will be used to assess the sense of vibration. The test will be applied to the first metatarsal head, medial foot, lateral foot and heel. The right and left extremities will be evaluated separately.

Discriminator (Baseline ® Discrimin-A-Gon 2) for the assessment of the sense of two-point separation- Point Discriminator, New York, USA) will be used. The test will be applied to the first metatarsal head, medial foot, lateral foot and heel.The right and left extremities will be evaluated separately.

For balance and walking; Tinetti Balance and Walking Test will be applied. Reaction time will be assessed by the Nelson foot test. By taking five measurements, the best and worst values will be discarded, and the average of the remaining three measurements will be recorded as the distance at which the ruler fell.

ELIGIBILITY:
Inclusion Criteria:

1. To be male and between the ages of 18-65,
2. For the study group, diagnosed with opioid use disorder according to the diagnostic criteria of the Diagnostic and Statistical Manual of Mental Disorders V (DSM V) and being on maintenance treatment,
3. To voluntarily agree to participate in the study,

Exclusion Criteria:

1. Having any systemic or neurological disease,
2. To have a cognitive effect at a level that will affect communication,

Ages: 18 Years to 65 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — Males
Study Population: This study will be conducted with the participation of 138 individuals, 40 individuals and 40 healthy individuals, between the ages of 18-65, who voluntarily agreed to participate in the study, who had an opioid use disorder according to DSM V diagnostic criteria and who were in the process of maintenance treatment.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-24 (Estimated)

PRIMARY OUTCOMES:
Plantar sensation -Tactile sense- | 1. Day
  Tactile sense was assessed using a full Semmes-Weinstein Monofilament test kit (North Coast Medical, San Jose, CA, USA). The smallest (1.65) monofilament was used firstly. The trial test was performed once before the assessment with eyes open and closed to introduce the test to each child. The monofilament was held perpendicular to the skin and pressed into the skin until it was slightly dished and held for 1.5 s in the pressed region and 1.5 s in the air. The child was asked to indicate if he/she felt the touch.
Plantar sensation - Vibration sense- | 1. Day
  A 128 Hz tuning fork (Baseline® Tuning Fork, New York, USA) was used to assess the vibration sense. The duration of the vibration was measured by a chronometer, started when the fork touched to the child's skin and stopped when the child indicated that "it has finished".
Plantar sensation - Two-point discrimination sense- | 1. Day
  A discriminator (Baseline®Discrim-A-Gon 2-Point Discriminator, New York, USA) was used for the assessment of the two-point discrimination sense. The assessment was started at the maximum distance and gradually decreased until the child was not able to differentiate the two points. When the subject felt the two points as one in two of the three trials, the distance was noted in mm. Light pressure was applied simultaneously at both ends of the discriminator to apply as equal pressure as possible.
Reaction time - Foot reaction time- | 1. Day
  Reaction time was evaluated with Nelson's foot test. For the test, the subject sits against the wall with the toe tip 2.5 cm and the heel part 5 cm. The test administrator will hold the reaction ruler between the wall and the subject's foot, and when the subject is ready, he will release the ruler and the subject holds the fallen ruler by squeezing it against the wall with his foot. Five measurements were taken and the best and worst values were discarded, and the average of the remaining three measurements was recorded as the distance the ruler fell.
Proprioception-Neck proprioception | 1. Day
  For neck prorioception; One end of the dual digital inclinometer is placed at the level of the 7th cervical vertebra and the other end is placed on the apex of the participant's head. The person is asked to close their eyes. After the neck is brought to the reference angle, it is ensured that the person perceives the angle by waiting for 10 seconds. Then, the person is asked to bring his head to an upright position and then repeat the taught reference angle as he perceives it. The absolute value of the angle at which it deviates from the target is recorded. In our study, 30° neck flexion will be accepted as the target angle value and the average of the evaluations was taken by making 3 evaluations.
Proprioception-Trunk proprioception | 1. Day
  For trunk proprioception, in the standing position, the first part of the inclinometer is fixed on the S1 spinous process, which is located and marked by palpation, and the second part is fixed on the T1 spinous process, which is also determined and marked by palpation, and the eyes of the person are closed. After the body is brought to the reference angle, it is ensured that the person perceives the angle by waiting for 10 seconds. Then, the person is asked to bring his/her torso to an upright position and then repeat the taught reference angle as he/she perceives it. The absolute value of the angle at which it deviates from the target is recorded. In our study, 30° trunk flexion will be accepted as the target angle value, and 3 evaluations were made and the average of the evaluations was taken.
Posture | 1. Day
  Posture assessment was done with the New York Posture Analysis (NYPA). The NYPA is a quantitative scale that evaluates whether the alignment of various body segments is appropriate for an individual in an anatomical position. NYPA has a form in which the body is examined in thirteen separate sections, and the posture assessment is scored using the visuals in these sections.
Balance and Gait-Tinetti Balance And Gait Test | 1. Day
  For balance and walking; Tinetti Balance and Gait Test was applied. The balance test includes sitting balance, standing and standing balance, evaluation of balance with eyes open and closed, 360 degree rotation around itself and evaluation of reaching. In the walking test, initiation of walking, step height, step width, step symmetry, step continuity, deviation from the walking line and trunk stability are evaluated. The questions are scored between 0-2, with a maximum of 26 points for balance and a maximum of 9 points for walking, with a total maximum score of 35. A total score of 18 or less indicates a high risk of falling, a score of 19-24 indicates a moderate fall risk, and a score of 24 and above indicates a low risk of falling.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided